CLINICAL TRIAL: NCT01057004
Title: EVIdence Based TreAtment - Heart Failure (EVITA-HF)
Acronym: EVITA-HF
Status: Completed | Type: Observational
Sponsor: Stiftung Institut fuer Herzinfarktforschung (Other)
Collaborators: Vifor Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: EVITA-HF
Record Dates: First submitted 2010-01-26; First posted 2010-01-27 (Estimated); Last update posted 2016-06-24 (Estimated); Status verified 2016-06

CONDITIONS: Heart Failure
Keywords: heart failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- all patients: chronical heart failure and EF ≤ 40 %

SUMMARY:
EVITA should function as an idea supplier and should coordinate possible future studies. Other important tasks of the register are: (i) the establishment of recommendations for an optimal medicinal therapy (OMT) as well as for ICD- and CRT-treatment; (ii) the establishment of quality assurance measures, including monitoring of new therapy.

DETAILED DESCRIPTION:
Cardiac insufficiency is the main or secondary diagnosis of 10% of all hospitalised patients. Due to the age-structure of the population and to the increased life expectancy after myocardial infarction prevalence is increasing. Even though prognosis in patients with established heart failure has been improved it remains serious, with an average survival rate of 50% after 4 years. Approximately 2% of all expenses in health care are caused by cardiac insufficiency, the most expensive being the hospitalization phase. The rehospitalisation rate after the first hospital stay is 50% within 6 months. By optimal, guideline-adjusted therapy during hospital- and post-hospital-stay the rehospitalisation rate could be reduced by 50%.

But our knowledge concerning therapies is based on study results, which are generated with selected patients under controlled study conditions. Thus it is necessary to collect data on the development of therapy, the successes as well as the complications in clinical everyday life. Results concerning the quality of therapies are required and measures are needed that will contribute to quality assurance and improvement. Due to these reasons EVITA was initiated with the following objectives, aims, structure, and organization form:

The register will not substitute randomized, controlled, multi-center clinical trials (RCT) that have a defined prospective research question. Such randomized studies investigate the "efficacy" of a therapy, i.e. a clinical effect under experimental conditions. In contrast, registers investigate the transferability of RCT results to the daily routine within hospital, the so called "effectiveness". Both study types are complementary and are needed for a judgment of the clinical efficiency as well as of security aspects and possible adverse reactions. Furthermore EVITA should function as an idea supplier and should coordinate possible future studies. Other important tasks of the register are: (i) the establishment of recommendations for an optimal medicinal therapy (OMT) as well as for ICD- and CRT-treatment; (ii) the establishment of quality assurance measures, including monitoring of new therapy. Every 6 months each study center receives a complete overview concerning the centers own data in comparison with the data supplied by other centers.

ELIGIBILITY:
Inclusion Criteria:

* chronical heart failure
* EF ≤ 40 %

Exclusion Criteria:

* no informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 4560 (Actual)
Dates: Start 2009-02; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Characteristics of consecutive patients with chronic cardiac insufficiency and an EF ≤ 40% in hospital daily routine within Germany | Admission to Hospital and 12 months thereafter

SECONDARY OUTCOMES:
Specification of the medical therapy according to the guidelines | Admission to hospital and 12 months thereafter
Monitoring of innovations of new therapy possibilities once these are introduced on the market | Admission to Hospital and 12 months thereafter
Specifications of implantable devices including ICD and CRT as well as the procedure of implantation and the success of the surgical intervention | Admission to Hospital and 12 months thereafter
Further interventions during clinical stay, after the index-event | Index hospital stay
Hospital mortality and non-fatal complications | Index hospital stay
Mortality and non-fatal complications within the first year | Admission to Hospital and 12 months thereafter
Symptomatic and frequency of rehospitalisation | Discharge after index hospital stay and 12 months thereafter
Medicinal and non-medicinal therapy after 12 months | 12 months after index hospital stay
Association between iron therapy and prognosis in patients with heart failure | Hospital admission and 12 months thereafter
  Analysis of laboratory values of hemoglobin, erythrocytes, reticulocytes, ferritin, serum iron, transferrin, transferrin saturation and their effect on prognosis of heartfailure patients. (RAID-HF substudy to EVITA-HF registry)

CONTACTS AND LOCATIONS:
Overall Officials: Jochen Senges, MD, Principal Investigator — Stiftung Institut für Herzinfarktforschung
Locations (11):
- Germany (11):
  - Universitätsklinikum Heidelberg, Heidelberg, Baden-Wurttemberg
  - Zentralklinikum Augsburg, Augsburg, Bavaria
  - Klinikum Coburg, Coburg, Bavaria
  - Klinikum Nürnberg, Nuremberg, Bavaria
  - Universitätsklinikum Würzburg, Würzburg, Bavaria
  - Klinikum Links der Weser Bremen, Bremen, City state Bremen
  - Universitätsklinik Rostock, Rostock, Mecklenburg-Vorpommern
  - Klinikum Lippe-Detmold, Detmold, North Rhine-Westphalia
  - Universitätsklinikum Essen (Klinik für Kardiologie), Essen, North Rhine-Westphalia
  - Elisabeth - Krankenhaus (Kardiologie) Essen, Essen, North Rhine-Westphalia
  - Universitätsklinikum des Saarlandes, Homburg/Saar, Saarland

IPD SHARING:
Plan to Share IPD: No